CLINICAL TRIAL: NCT04748081
Title: Evaluation of the Bleeding Risk Associated With Hepatectomy: a Nationwide Population-based Study
Brief Title: The Major Bleeding Risk Following Hepatectomy
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: An-Nan Hospital, China Medical University (Other); Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: CMUH104-REC2-115
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Gastrointestinal Hemorrhage; Postoperative Hemorrhage; Surgery--Complications
Keywords: Gastrointestinal hemorrhage; Hepatectomy; Postoperative hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Postoperative Hemorrhage | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery cohort: Patients who underwent hepatectomy (ICD-9-CM procedure code: 50.2, 50.22, 50.3 and 50.4) between 2000 and 2012 were identified as the surgery cohort.
  Interventions: Procedure: hepatectomy
- Control cohort: Patients without any record of hepatectomy between 2000 and 2012 were defined as the control cohort.

INTERVENTIONS:
Procedure: hepatectomy — hepatectomy (ICD-9-CM procedure code: 50.2, 50.22, 50.3 and 50.4)
  Groups: Surgery cohort

SUMMARY:
This study examined long-term incidence rates of major bleeding associated with hepatectomy. The investigators used data from Taiwan's National Health Insurance Research Database. Patients who underwent hepatectomy between 2000 and 2012 were identified by International Classification of Diseases, Ninth Revision, Clinical Modification codes. Variables including gender, age, comorbidities, and prescribed medications were matched between cases and controls. A total of 1,053 patients with hepatectomy and 4,212 matched non-hepatectomy subjects were included in this study.

DETAILED DESCRIPTION:
The study population consisted of two cohorts. Patients who underwent hepatectomy (ICD-9-CM procedure code: 50.2, 50.22, 50.3 and 50.4) between 2000 and 2012 were identified as the surgery cohort. The index date was defined as the earliest date that patients underwent hepatectomy. Patients without any record of hepatectomy during the same period of time were defined as the control cohort. Patients younger than 20 years of age and those diagnosed with coagulation defects (ICD-9-CM: 286.4) or had a pre-existing bleeding episode before the index date. The primary outcome of this study was an incident diagnosis of major bleeding, consisting of 3 categories: intracranial bleeding (ICD-9-CM; 430, 431, 432.0, 432.1, 432.9, 852.0, 852.2, 852.4, 853.0), gastrointestinal (GI) bleeding (ICD-9-CM; 456.0, 456.20, 530.7, 531, 531.2, 531.4, 531.6, 532, 532.2, 532.4, 532.6, 533, 533.2, 533.4, 533.6, 534, 534.2, 534.4, 534.6, 535.01, 535.11, 535.21, 535.31, 535.41, 535.51, 535.61, 535.71, 537.83, 537.84, 562.02, 562.03, 562.12, 562.13, 569.3, 569.85, 578) and other sites bleeding [ICD-9-CM; 336.1, 363.6, 372.72, 376.32, 377.42, 379.23 (eye); 593.81, 866.01, 866.02, 866.11, 866.12 (kidney); 719.1 (joint); 729.92 (soft tissue); 423.0 (heart); 772.5 (adrenal gland), 626.8, 626.9 (uterine)].

Demographic characteristics evaluated in this study included gender, age, comorbidities and prescribed medications. The comorbidities included hypertension (ICD-9-CM; 401-405, A260 and A269), hyperlipidemia (ICD-9-CM: 272), chronic liver disease (ICD-9-CM: 571.4, 571.5), hepatitis C virus (HCV) infection (ICD-9-CM: 070.41, 070.44, 070.51, 070.54, and V02.62), malignant neoplasm of liver and intrahepatic bile ducts (ICD-9-CM: 155), cirrhosis (ICD-9-CM: 571, A347), chronic kidney disease (ICD-9-CM: 580-589, A350), alcohol-related disease (ICD-9-CM: 291, 303, 305.0, 357.5, 425.5, 535.3, 571.0-571.3, 980.0, E947.3), biliary stone disease (ICD-9-CM: 574), and diabetes mellitus (ICD-9-CM: 250). The investigators also searched the clinical records for the use of anticoagulants, antiplatelets, thrombolytic agents, non-steroidal anti-inflammatory drugs (NSAIDs), serotonin-norepinephrine reuptake inhibitors (SNRIs) and selective serotonin reuptake inhibitors (SSRIs) prescribed before the index date. The investigators applied a 4:1 propensity-score matched analysis to reduce selection bias between cases and controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent hepatectomy between 2000 and 2012.

Exclusion Criteria:

* Patients younger than 20 years of age
* Patients diagnosed with coagulation defects or had a pre-existing bleeding episode before the earliest date that patients underwent hepatectomy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent hepatectomy (ICD-9-CM procedure code: 50.2, 50.22, 50.3 and 50.4) between 2000 and 2012, and without past history of coagulation defects and bleeding episodes.
Sampling Method: Probability Sample
Enrollment: 5265 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incident diagnosis of major bleeding | From the the earliest date that patients underwent hepatectomy to the date of an incident diagnosis of major bleeding, December 31, 2015 or withdraw from National Health Insurance Research Database (NHIRD).
  Major bleeding consists of 3 categories: intracranial bleeding (ICD-9-CM; 430, 431, 432.0, 432.1, 432.9, 852.0, 852.2, 852.4, 853.0), gastrointestinal (GI) bleeding (ICD-9-CM; 456.0, 456.20, 530.7, 531, 531.2, 531.4, 531.6, 532, 532.2, 532.4, 532.6, 533, 533.2, 533.4, 533.6, 534, 534.2, 534.4, 534.6, 535.01, 535.11, 535.21, 535.31, 535.41, 535.51, 535.61, 535.71, 537.83, 537.84, 562.02, 562.03, 562.12, 562.13, 569.3, 569.85, 578) and other sites bleeding [ICD-9-CM; 336.1, 363.6, 372.72, 376.32, 377.42, 379.23 (eye); 593.81, 866.01, 866.02, 866.11, 866.12 (kidney); 719.1 (joint); 729.92 (soft tissue); 423.0 (heart); 772.5 (adrenal gland), 626.8, 626.9 (uterine)].

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No